CLINICAL TRIAL: NCT00995696
Title: Pharmaceutical Safety Tracking (PhaST): Managing Medications for Patient Safety
Brief Title: Treatment Follow-up Study
Acronym: PhaST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: William Gardner, PhD, The Research Institute at Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 11062007; 5R18HS017258 (AHRQ)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Interactive Voice Response (IVR)
Keywords: Interactive Voice Response (IVR); Antidepressant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PhaST (Experimental): Group receiving PhaST IVR phone calls.
  Interventions: Behavioral: PhaST IVR Calls
- Usual Care (No Intervention): Group NOT receiving IVR phone calls.

INTERVENTIONS:
Behavioral: PhaST IVR Calls — Participants in this condition receive 7 computer automated IVR calls.
  Arms: PhaST

SUMMARY:
This study will assess the effectiveness of a medication safety monitoring method utilizing interactive voice response technology for youth recently prescribed anti-depressant medication.

DETAILED DESCRIPTION:
Over a two year period, 800 children and adolescents between the ages of 6 - 17 years old who have received a new prescription for an antidepressant will be recruited from families receiving care at Nationwide Children's Hospital or Community Physician Practices affiliated with Nationwide Children's Hospital.

At the baseline site visit, a research assistant will explain the study to the family and obtain written informed consent from the subject's parent/guardian and assent from the youth. In addition, consent for release of information will be obtained from the parent/guardian to communicate with the treating physician and other professionals involved in the youth's mental health care (if applicable) as well as to obtain medical records. Randomization to study condition will also be conducted by this RA and a description of the PhaST procedure will be given to the families randomized into that condition.

Once informed consent and assent has been obtained, a second research assistant will administer our assessment battery to the family. This RA will serve as an independent research evaluator and will determine whether the patient has experienced an adverse event during the past month. A comprehensive assessment of adverse events will be conducted with individuals at study entry (baseline) and once a month following for three months. At each assessment, the primary parent informant and child will be interviewed separately and concurrently.

For patients in the PhaST condition, PhaST will monitor the patient through a series of brief telephone calls following the FDA's recommendations for frequency of visits. There will be a total of seven calls over the same three-month period as the visits. The first four calls will be weekly. The next two calls will be every two weeks. The final call will be one month later. The monitoring call presents the 8-question PhaST screening assessment and lasts an average of only 2 minutes and 12 seconds. To ensure that the health data are secure, the patients or parents identify themselves with PINs at the beginning of an automated call. Parents answer the questions for children 12 years old or younger and teenagers answer for themselves. If a patient answers "no" to all the screening questions, the data are automatically stored and a report is routed to the patient's electronic health record and to the patient's clinician's electronic inbox. If a patient answers "yes" to any screening questions, the on-call PTS will immediately be paged.

For any "yes" responses to a screening question, the PTS will follow-up and triage the severity of the problem using a semi-structured clinical interview. Based on the triage interview, the PTS decides whether action is warranted. If the screen is a false positive (meaning, no adverse event is occurring), the PTS logs the data to be included in a report sent to the patient's psychiatrist and clinician (if applicable). If she judges that the case requires further attention, she will talk with parent(s)/ guardian(s) and patient regarding the development of plan to address potential risk. If the youth has a developed safety plan, she will review the plan with the family and talk with them about implementing or modifying the plan to address any potential risk.

If the PTS concludes that the case requires immediate further assessment, she will attempt to contact Nationwide Children's Hospital Psychiatry Consultation Service. If the psychiatrist on-call is not available and the child has a safety plan, the ongoing or on-call behavioral health provider(s) reflected in the safety plan will be contacted. If the professionals reflected in the safety plan are not available or the child does not have a safety plan, the Nationwide Children's Behavioral Health Crisis Team will be contacted. The professional who is reached by the PTS regarding the potential risk is responsible for managing the crisis.

ELIGIBILITY:
Inclusion Criteria:

* Over a two year period, 800 children and adolescents aged 6 - 17 years old who have received a new prescription for an antidepressant will be recruited from families receiving care at Nationwide Children's Hospital or Community Physician Practices affiliated with Nationwide Children's Hospital. It should be noted that we are not requiring this to be the first antidepressant prescription a patient has received.

Exclusion Criteria:

* Families who speak do not speak English and families with children who are actively psychotic.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Does the PhaST intervention increase the information in the clinical record systems about the patient's mental health during the follow-up period? | 3 months

SECONDARY OUTCOMES:
The investigators predict that PhaST patients will have a greater proportion of their recommended monitoring contacts. | 3 months
The investigators predict higher agreement between chart-documented adverse events and examiner-determined adverse events in the PhaST condition. | 3 months
The investigators predict that PhaST patients will have better medication adherence (a greater percentage of time with medication coverage) compared to Usual Care. | 3 months
The investigators predict parents will be more satisfied with care and report higher perceived child safety with PhaST versus Usual Care. | 3 months
The investigators predict that PhaST patients will have fewer depressive and anxiety symptoms, the primary targets of antidepressant drugs, than those in Usual Care. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William Gardner, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio